CLINICAL TRIAL: NCT01572168
Title: A Phase II Study of Acupuncture for the Treatment of Cancer Related Fatigue in Children and Adolescents With Central Nervous System Tumors
Brief Title: Acupuncture for the Treatment of Cancer Related Fatigue
Status: Terminated | Phase: Phase 2 | Type: Interventional
Why Stopped: slow accrual
Sponsor: Ann & Robert H Lurie Children's Hospital of Chicago (Other)
Responsible Party: Principal Investigator, Rishi Lulla, Prinicipal Investigator, Ann & Robert H Lurie Children's Hospital of Chicago
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Supportive Care
Other Study IDs: 2011-14423
Record Dates: First submitted 2012-02-24; First posted 2012-04-06 (Estimated); Last update posted 2016-02-05 (Estimated); Status verified 2016-02

CONDITIONS: Fatigue
Keywords: Fatigue
MeSH Terms: conditions — Fatigue | interventions — Acupuncture Therapy

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- Acupuncture (Experimental): Eight sessions of weekly acupuncture
  Interventions: Other: Acupuncture

INTERVENTIONS:
Other: Acupuncture — Eight session of weekly acupuncture

SUMMARY:
Cancer-related fatigue occurs in both adult and pediatric patients undergoing chemotherapy and/or radiation. Recently, methods to measure fatigue have improved - however, no non-medication interventions have been studied. Ameliorating fatigue may result in an improved quality of life for patients. Acupuncture is a safe and well-tolerated procedure and has been used for many indications in pediatric patients. Adult studies have suggested improvement in cancer-related fatigue after acupuncture in adults. In this trial, we propose using acupuncture for the treatment in cancer-related fatigue in children and adolescents with central nervous system tumors.

ELIGIBILITY:
Inclusion Criteria:

* Patients who are ≥ 8 year of age and ≤ 21 years of age who are undergoing chemotherapy and/or radiation therapy for the treatment of any primary or recurrent central nervous system tumor (regardless of diagnosis or disease stage, whether it is malignant or benign, and in any location) at Children's Memorial Hospital.
* Patients who recently completed therapy (within 60 days of enrollment) will also be eligible. Patients must have a minimum baseline fatigue score of 15 on the pedsFACIT-F scale (Range 0-44). This is not a standard assessment for required clinical care and will only be administered by a research assistant to any patient after consent has been obtained. The assessment will be done during a routine clinic visit.
* For patients receiving cytotoxic chemotherapy with a history of myelosuppression or radiation, a hemoglobin concentration of >8 g/dL measured within 10 days of enrollment and a platelet count of > 30,000 within 5 days of enrollment is required.
* Patients must also be able to read and understand English and read a computer screen.
* Patients with no known contraindications to acupuncture therapy.
* Patients who are able to attend all scheduled visits for acupuncture.
* Patients must have a Karnofsky Performance Score of ≥ 50% or a Lansky Performance Score of ≥ 50.
* Patients who have provided informed consent for the research study (parental consent for patients < 18 years of age). Patients between 12 years and 18 years of age must provide assent in additional to parental consents.

Exclusion Criteria:

* Patients with evidence of any cognitive dysfunction that would limit their abilities to report fatigue.
* Patients who have received acupuncture in the previous six weeks.
* Patients with a life expectancy < 3 months.
* Patients who are pregnant or lactating.
* Patients with a past history of therapy or scheduled visits non-compliance, as determined by their treating physician.

Ages: 8 Years to 21 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child, Adult
Enrollment: 7 (Actual)
Dates: Start 2011-09; Primary Completion 2015-12 (Actual); Study Completion 2015-12 (Actual)

PRIMARY OUTCOMES:
cancer-related fatigue | Participants will be on-study for up to 14 weeks. . No follow-up will be required after the completion of the study.

CONTACTS AND LOCATIONS:
Overall Officials: Rishi Lilla, MD, Principal Investigator — Ann & Robert H Lurie Children's Hospital of Chicago
Locations (1):
- Ann & Robert H. Lurie Children's Hospital of Chicago, Chicago, Illinois, United States

REFERENCES:
- [Background] Cella D, Davis K, Breitbart W, Curt G; Fatigue Coalition. Cancer-related fatigue: prevalence of proposed diagnostic criteria in a United States sample of cancer survivors. J Clin Oncol. 2001 Jul 15;19(14):3385-91. doi: 10.1200/JCO.2001.19.14.3385. PMID 11454886
- [Background] Lai JS, Cella D, Kupst MJ, Holm S, Kelly ME, Bode RK, Goldman S. Measuring fatigue for children with cancer: development and validation of the pediatric Functional Assessment of Chronic Illness Therapy-Fatigue (pedsFACIT-F). J Pediatr Hematol Oncol. 2007 Jul;29(7):471-9. doi: 10.1097/MPH.0b013e318095057a. PMID 17609625
- [Background] Libonate J, Evans S, Tsao JC. Efficacy of acupuncture for health conditions in children: a review. ScientificWorldJournal. 2008 Jul 13;8:670-82. doi: 10.1100/tsw.2008.86. PMID 18661055
- [Background] Jindal V, Ge A, Mansky PJ. Safety and efficacy of acupuncture in children: a review of the evidence. J Pediatr Hematol Oncol. 2008 Jun;30(6):431-42. doi: 10.1097/MPH.0b013e318165b2cc. PMID 18525459
- [Background] Molassiotis A, Sylt P, Diggins H. The management of cancer-related fatigue after chemotherapy with acupuncture and acupressure: a randomised controlled trial. Complement Ther Med. 2007 Dec;15(4):228-37. doi: 10.1016/j.ctim.2006.09.009. Epub 2006 Nov 13. PMID 18054724
- [Background] Balk J, Day R, Rosenzweig M, Beriwal S. Pilot, randomized, modified, double-blind, placebo-controlled trial of acupuncture for cancer-related fatigue. J Soc Integr Oncol. 2009 Winter;7(1):4-11. PMID 19476729
- [Background] Matecki, A.a.I., David, Acupunture for the Treatment of Chronic Post-Chemotherapy Fatigue. ClinicalTrials.gov, 2008: p. NCT00658034.